CLINICAL TRIAL: NCT06390176
Title: Lactobacillus Rhamnosus LGG Alleviates Oral Mucositis in Patients Undergoing Radiotherapy for Malignant Head and Neck Tumors: A Randomized Controlled Trial
Brief Title: Lactobacillus Rhamnosus GG Alleviates Oral Mucositis in Patients Undergoing Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-1747
Record Dates: First submitted 2024-04-21; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Placebo-containing tablets
  Interventions: Dietary Supplement: Placebo-containing tablets; Radiation: Radiotherapy
- Experimental group (Experimental): Lactobacillus rhamnosus GG (LGG)
  Interventions: Dietary Supplement: Lactobacillus rhamnosus GG powder; Radiation: Radiotherapy

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus GG powder — Lactobacillus rhamnosus GG powder (PROBIOTICS Powder, USA) contained no less than 5×10^8 CFU viable cells of Lactobacillus rhamnosus GG as the active ingredient.
  Arms: Experimental group
Dietary Supplement: Placebo-containing tablets — Starch preparations that look and taste like Lactobacillus rhamnosus GG powder
  Arms: Control group
Radiation: Radiotherapy — One of the inclusion criteria for the study was that patients with squamous carcinoma of the head and neck (including nasopharyngeal carcinoma) needed to receive either radiotherapy alone or simultaneous radiotherapy and chemotherapy, with radiotherapy using intensity-modulated radiotherapy techniques.

SUMMARY:
Radiation therapy is a common treatment modality in the management of head and neck malignancies. However, head and neck tumors often have some adverse reactions when receiving radiation therapy, such as dry mouth, change of taste, oral mucositis, etc. Among them, the incidence of oral mucositis is more than 90%, and the incidence of oral mucositis of degree 3 or more than degree 3 is more than 50%. Severe oral mucositis seriously affects the quality of survival of patients.

Lactobacillus rhamnosus GG (LGG) is a type of lactic acid bacterium, which is an important component of the microbiota in many parts of the human body.

Lactobacillus rhamnosus GG (LGG) is a lactic acid bacterium found in the human body, extensively researched for its probiotic properties. It has been tested in clinical trials for preventing and treating oral mucosal reactions during intensified radiotherapy for head and neck squamous cell carcinoma. LGG adheres well to epithelial layers, produces a protective biofilm, and modulates immune responses. It shows promise in reducing radiation-induced oral mucositis and can be safely used in infant formula. Additionally, a daily dosage of 3×10^9 CFU of LGG has been effective in treating irritable bowel syndrome without adverse effects

DETAILED DESCRIPTION:
Radiotherapy (RT) is an important treatment for head and neck malignant tumors and can be used alone or in combination with chemotherapy as radical or adjuvant therapy. Despite improvements in RT equipment and techniques, there are still a variety of acute oral complications, including oral mucositis (OM), xerostomia, taste dysfunction, and oral infection. OM is one of the most common acute radiation-related toxicity in head and neck malignant tumor patients receiving RT, and approximately 50~70% of patients experience severe oral mucositis (SOM). The painful inflammation and ulceration associated with OM not only profoundly affect patients' ability to eat, swallow, and speak but also decrease patients' tolerance to anti-cancer treatment, seriously impairing patients' quality of life (QoL) and causing interruptions and cancellations of cancer treatment. Standard treatment for OM focuses on pain control, rehydration, and good oral hygiene. For patients with hematopoietic stem cell transplantation, palifermin (keratinocyte growth factor-1) is recommended. Although some clinical strategies for OM such as non-steroidal anti-inflammatory drugs, mucosal protective agents, growth factors and cytokines, antibacterial, and pain relief drugs have been recommended by the Multinational Association of Supportive Care in Cancer and International Society of Oral Oncology (MASCC/ISOO), the therapeutic benefit is limited6. Thus, it is crucial to develop effective drugs or treatment strategies to decrease radiation-induced mucosal toxicity.

LGG has been used in clinical trials for the prevention and treatment of oral mucosal reactions during intensified radiotherapy for head and neck squamous cell carcinoma (including nasopharyngeal carcinoma). It was isolated from a healthy adult's fecal sample and possesses good growth characteristics and the ability to adhere to epithelial layers. It has long been one of the most extensively researched and applied probiotic strains, utilized in various commercially available probiotic products. Its beneficial effects have been extensively studied in clinical trials and human intervention studies, including its role in preventing and treating gastrointestinal infections and diarrhea, stimulating immune responses, and even preventing certain allergic symptoms.

In addition to producing a biofilm that mechanically protects the mucosa, reduces epithelial cell apoptosis, and maintains cell cytoskeleton integrity, LGG also exhibits immunomodulatory properties. It protects the epithelium from radiation damage by reducing TLR-2/COX-2 activation and regulates the protein levels of pro-inflammatory cytokines tumor necrosis factor-alpha, interleukin-6, and monocyte chemotactic protein-1 in tissues, actively participating in host defense processes. It can also reduce the number of pathogenic bacteria and regulate colony distribution.

The occurrence and development of radiation-induced oral mucositis are closely related to cellular immunity. A series of pro-inflammatory cytokines produced by immune cells such as tumor necrosis factor-alpha and interleukin-6 will positively feedback to amplify the inflammatory response of radiation-induced oral mucositis.

Regarding safety, LGG can be added to infant formula as a probiotic. Furthermore, studies have shown that a dosage of 3×10^9 CFU of LGG per day can be used to treat irritable bowel syndrome (IBS) without causing disease or toxicity in the body. Therefore, Lactobacillus rhamnosus GG holds promise as a potential approach for preventing and treating radiation-induced oral mucositis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients pathologically diagnosed with non-metastatic head and neck malignant tumors;
2. Aged 18-80 years;
3. Eastern Cooperative Oncology Group performance status of ≤2;
4. Planning to receive definitive RT or postoperative adjuvant RT;
5. Normal liver, kidney and bone marrow function;
6. Sign informed consent.

Exclusion Criteria:

1. Known hypersensitivity or more severe allergies to Lactobacillus Reuteri components;
2. Those with poor compliance;
3. Pregnancy or breastfeeding;
4. History of head and neck radiotherapy;
5. Taking antifungal or viral medications one week prior to the start of radiation therapy.
6. Other patients (with any other serious other medical condition) who, in the opinion of the investigator, are not suitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale.The WHO Oral Toxicity Scale categorizes oral mucositis into grades 0-4, with the higher the grade the more severe the patient's oral mucositis. Grade 0 means that the oral mucosa is normal and the patient has no symptoms or signs; grade 1 means that the mucosa is erythematous with or without pain and does not interfere with eating; grade 2 means that the mucosa is erythematous and ulcerated, but still able to eat solid food; grade 3 means that the mucosa is severely ulcerated with extensive erythema and unable to eat solid food; and grade 4 means that the ulcers of the mucosa are fused together into a sheet, and their severity is so severe that it is not possible to eat.

SECONDARY OUTCOMES:
The time to onset of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  Time from the first day of radiotherapy to the first determination of SOM. Patients without observed SOM were assigned onset days of 6 or 6.5 weeks
The duration of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  The first determination of SOM to the first instance of non-severe OM (WHO grade <3), without a subsequent instance of SOM. Patients without observed SOM were assigned a duration of 0 days
Xerostomia summated xerostomia inventory (SXI) | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  Xerostomia is subjectively assessed on the Summated Xerostomia Inventory (SXI). The SXI is categorized according to score as 0 no dry mouth (5), 1 mild dry mouth (6-8), 2 moderate dry mouth (9-12), and 3 severe (13-15). Objectively the researchers measured the salivary flow rate to rate dry mouth, i.e., a 2% citric acid solution was applied to the side of the tongue every 30 seconds for 5 minutes, the secreted saliva was flowed into a sterile tube and the salivary flow rate (ml/min) was calculated, normal stimulated salivary flow rate was between 1.5 - 2.0 mL/min and low stimulated salivary flow rate was < 0.5 ~ 0.7 mL/min.
Functional assessment of cancer therapy-head and neck (FACT- H&N) quality of life questionnaire | 1 week before radiotherapy; at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); ; and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  FACT- H&N quality of life questionnaire 4.0 is a scale used to assess quality of life in patients with head and neck tumors. It includes all aspects of quality of life, such as physical, emotional, functional, and social. With this scale, physicians can gain a more comprehensive understanding of a patient's quality of life status, which can lead to better treatment planning and support. The FACT-HN 4.0 scale has a total score range of 0-180, which includes four dimensions such as physical health, social/family, emotional, and functional/symptomatic. Each dimension has a different range of scores.The lowest score is 0, which indicates the worst quality of survival, and the highest score is 180, which indicates the best quality of survival. As the score increases, it indicates a better quality of survival; conversely, as the score decreases, it indicates a decreased quality of survival.
Adverse events | From the first day of radiotherapy to the day of the last radiation dose received, usually 6 or 6.5 weeks
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version
Oral activities scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy. The evaluation period is approximately 6 weeks and 6 1/2 weeks
  Patients report the degree to the impact of MTS on oral activities (including swallowing, drinking, eating, talking, sleeping) (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms
Mouth and throat soreness (MTS) scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6 1/2 weeks
  Patients report mouth and throat soreness (MTS) scores (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No